CLINICAL TRIAL: NCT01809301
Title: A Single-Dose, Randomized, Open-Label, Crossover, Comparative Bioavailability Study of TRIA-662 500 mg Immediate-Release Tablets and NIASPAN 1000 mg Extended-Release Tablets in Healthy Male and Female Volunteers Under Fed Conditions
Brief Title: Comparison of TRIA-662 500 mg and Niaspan 1000 mg in Healthy Male and Female Volunteers Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortria Corporation (Industry)
Collaborators: PPD Development, LP (Industry); Pharmena North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BPSI-1479
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
Keywords: Bioavailability
MeSH Terms: interventions — Niacin; N(1)-methylnicotinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Niaspan (Active Comparator): Single dose of one NIASPAN® 1000 mg Extended-Release Tablet following dinner
  Interventions: Drug: Niaspan
- TRIA-662 (Experimental): Single dose of two TRIA-662, 500 mg Immediate-Release Tablets following dinner
  Interventions: Drug: TRIA-662

INTERVENTIONS:
Drug: Niaspan
  Other Names: Extended-release nicotinic acid; Extended-release niacin
  Arms: Niaspan
Drug: TRIA-662
  Other Names: 1-methynicotinamide chloride; N-methylnicotinamide chloride; MNA chloride; 1-MNA chloride
  Arms: TRIA-662

SUMMARY:
The objective of this study is to compare the absorption of a niacin metabolite (1-methylnicotinamide, 1-MNA) from TRIA-662 (1-methylnicotinamide chloride)relative to the production of 1-MNA from Niaspan. The 1-MNA information obtained from this study will be used to adjust the top dose of a planned TRIA-622 efficacy study.

ELIGIBILITY:
Main Inclusion Criteria

1. Healthy, non-smoking (for at least 6 months prior to drug administration), male and female volunteers, 35-65 years of age, inclusive.
2. Body weight within 30% of ideal body weight.
3. Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the Principal Investigator/Sub-Investigator.
4. Systolic blood pressure between 100-140 mmHg, inclusive, and diastolic blood pressure between 60-90 mmHg, inclusive, and heart rate between 50-100 bpm, inclusive, unless deemed otherwise by the Principal Investigator/Sub-Investigator.

Main Exclusion Criteria

1. Known history or presence of any clinically significant hepatic (e.g. active liver disease, hepatic necrosis, jaundice, hepatobiliary disease, hepatic dysfunction), renal/genitourinary (e.g. renal impairment, renal dysfunction), gastrointestinal, cardiovascular (e.g. angina, myocardial infarction), cerebrovascular, pulmonary, endocrine (e.g. diabetes, hypophosphatemia,), immunological, musculoskeletal (e.g. rhabdomyolysis, myopathy), neurological, psychiatric, dermatological or hematological or condition unless determined as not clinically significant by the Principal Investigator/Sub-Investigator.
2. Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first drug administration, as determined by the Principal Investigator/Sub-Investigator.
3. Known presence of active bleeding.
4. Known history or presence of:

   * Alcohol abuse or dependence within one year prior to drug administration.
   * Drug abuse or dependence.
   * Hypersensitivity or idiosyncratic reaction to niacin, its excipients (e.g. methyl cellulose, povidone, stearic acid), and/or related substances (e.g. nicotinamide [Vit. B3]).
   * Hypertension requiring treatment
   * Active peptic ulcer
   * Hypo or hyperthyroidism not treated or not stable for at least 6 months
   * Gout
   * Food allergies and/or presence of any dietary restrictions.
   * Severe allergic reactions (e.g. anaphylactic reactions, angioedema).
5. Intolerance to and/or difficulty with blood sampling through venipuncture.
6. Use of any prescription medication within 30 days prior to drug administration (except for hormonal contraceptives).
7. Use of any over-the-counter medications or vitamins (including herbal and/or dietary supplements and/or teas) within 14 days prior to drug administration (except for spermicidal/barrier contraceptive products).
8. Use of any statins (e.g. lovastatin, simvastatin), bile acid sequestrants (e.g. cholestyramine), aspirin, antihypertensive therapy, vasoactive drugs (e.g. nitrates), calcium channel blockers, adrenergic blocking agents, anticoagulants and vitamins (e.g. multivitamins) within 30 days prior to drug administration.
9. Women who are pregnant, planning to become pregnant during the study or are nursing.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
ANOVA and 90% Confidence Intervals on ln-transformed, baseline corrected molar urine recovery data of niacin metabolites. | 96 hours of urine collection

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax)of each niacin metabolite | Pre-dose and at 1, 2, 3, 5, 6, 12, 16, 20, 24 and 30 hours after dosing in each study period.
Plasma area under the curve to the last measureable timepoint, AUCt | Pre-dose and at 1, 2, 3, 5, 6, 12, 16, 20, 24 and 30 hours after dosing in each study period.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio A Cefali, PharmD, PhD., Study Chair — Cortria Corporation
Locations (1):
- Bio Pharma Services Inc. (BPSI), Toronto, Ontario, Canada